CLINICAL TRIAL: NCT02972021
Title: High Flow Nasal Cannulae Oxygen Therapy in Respiratory Insufficiency Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Chen Yuanzhuo, department of emergency, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: shsk20160722
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Patients With Respiratory Insufficiency
Keywords: respiratory insufficiency; High-flow nasal cannula
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Other): Pure oxygen by nasal cannula group
  Interventions: Device: High-flow nasal cannula
- HFNC (Experimental): oxygen by High-flow nasal cannula
  Interventions: Device: High-flow nasal cannula

INTERVENTIONS:
Device: High-flow nasal cannula

SUMMARY:
Chronic respiratory insufficiency in patients with advanced disease to the late treatment depends mainly on mechanical ventilation and other high intensity respiratory support therapy. Strengthen the stability of chronic respiratory insufficiency intervention can reduce the frequency and extent of acute disease, saving medical resources.High-flow nasal cannula (HFNC), as a new non-invasive oxygen therapy system, has gradually become a weapon of respiratory support therapy. There is little research on the role of HFNC in oxygen therapy for chronic respiratory insufficiency.

Our previous studies have found the potential value of HFNC in chronic respiratory insufficiency. The aim of this project is to promote the use of HFNC in the t reatment of chronic respiratory insufficiency in HFRS in Shanghai first, second and third grade hospitals in an effort to confirm that HFNC can improve the prognosis of patients with chronic respiratory insufficiency compared with nasal oxygen therapy.

DETAILED DESCRIPTION:
1. To confirm HFNC used in patients with chronic respiratory insufficiency oxygen therapy than the general nasal catheter oxygen and the difference between what better.
2. We set up a point of research in the tertiary hospitals, secondary hospitals and primary hospitals to explore the different levels of HFNC in the application of the efficacy of the hospital there are differences and what is better. To further clarify the promotion of HFNC to secondary hospitals and primary hospitals have no meaning.
3. Patients with chronic respiratory insufficiency who required long-term oxygen therapy were randomized to a randomized, controlled, multicentre clinical trial of HFNC with nasal oxygen therapy. Analysis and comparison of HFNC and general nasal catheter oxygen in the treatment of chronic respiratory insufficiency there is no difference, HFNC in different grades of hospital use is consistent.
4. Research methods:

4.1 Subjects: Chronic respiratory insufficiency required long-term oxygen therapy to Shanghai Tenth People's Hospital and multi-center hospital patients.

4.2 Study sample size: 100 samples were collected from each of the three test centers. Of which 150 cases of nasal oxygen therapy, HFNC 150 cases.

ELIGIBILITY:
Inclusion Criteria:

- Patients with chronic respiratory insufficiency who require long-term oxygen therapy.

Age 18-85 years old. Agree to participate in this study.

Exclusion Criteria:

- Patients with advanced respiratory support (invasive mechanical ventilation, noninvasive mechanical ventilation) indications Cardiovascular disease caused by respiratory insufficiency Immune dysfunction caused by respiratory insufficiency Tumor-induced respiratory insufficiency People with disturbance of consciousness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Improve dyspnea score | up to 12 months after oxygen therapy
Length of hospital stay | up to 12 months after oxygen therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth Hospital, Shanghai, Shanghai Municipality, China